CLINICAL TRIAL: NCT00091923
Title: A Randomized Trial to Evaluate 2 Hours of Daily Patching for Amblyopia in Children 3 to <7 Years Old
Brief Title: Trial to Evaluate 2 Hours of Daily Patching for Amblyopia in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEI-96; 2U10EY011751 (NIH); 5U10EY011751 (NIH)
Record Dates: First submitted 2004-09-20; First posted 2004-09-22 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2009-09

CONDITIONS: Amblyopia
MeSH Terms: conditions — Amblyopia | interventions — Eyeglasses

INTERVENTIONS:
Device: Eye patch
Device: Spectacles

SUMMARY:
The objectives of the Spectacle Phase are:

* In previously untreated pure anisometropic patients (i.e. patients who have not used spectacles in the last year and who do not have strabismus), to determine

  1. the incidence of resolution of amblyopia with spectacle correction alone and
  2. the time course of visual acuity improvement with spectacle correction alone.
* In all other patients, to achieve maximal improvement with spectacle correction prior to entering the randomized trial.

The objectives of the Randomized Trial are:

* To determine whether 5 weeks of patching treatment (2 hours of patching per day of the sound eye combined with at least one concurrent hour of near activities), compared with a control group (using spectacle correction only), improves visual acuity in patients with moderate to severe amblyopia (20/40 to 20/400).
* To determine the maximal improvement and time course of improvement with this patching treatment regimen.

DETAILED DESCRIPTION:
There are few data on the improvement that occurs with spectacle correction alone in cases of anisometropic amblyopia. The only published study of which we are aware is that of Moseley, et al, who found that 8 of 12 patients prescribed spectacles for the first time improved 3 or more lines in the amblyopic eye. Therefore, the Spectacle Phase of the current study will provide important information related to the management of patients with anisometropic amblyopia.

Additionally, despite clinical experience that strongly indicates that amblyopia can be improved with treatment, there are those who claim that the benefit of treatment is unproven. Although improvement with amblyopia therapy has been shown in prospective trials, there have been no conclusive data published from a randomized trial evaluating the effect of amblyopia treatment compared with a control group. Therefore, we have designed a randomized trial to definitively address this issue.

In the trial, the effect on amblyopic eye acuity after five weeks of 2 hours of prescribed daily patching (combined with at least one hour of concurrent near activities) will be compared with a control group using spectacle correction only. In a study conducted by the Pediatric Eye Disease Investigator Group, a 2-hour daily patching treatment regimen improved moderate amblyopia (20/40 to 20/80) by an amount similar to the improvement seen with 6 hours of daily patching.

At the end of five weeks, patients whose amblyopic eye has improved from baseline will continue in follow up, using the assigned treatment, until the amblyopic eye acuity stops improving or until the amblyopia resolves. This will provide data on the maximum improvement achievable with this treatment regimen and on the time course to reach maximal improvement. There is no known harm in deferring treatment of amblyopia for five weeks in the age range to be included in the trial (3 to <7 years old). Standard care for a patient with amblyopia includes prescribing spectacle correction and having the patient return in 4 to 6 weeks for measurement of visual acuity. Spectacles alone are continued as long as the acuity in the amblyopic eye is improving. Once the acuity stops improving, occlusion or other active treatment is initiated. The maximum delay in active treatment of the control group beyond the standard of care is 5 weeks. In our prior Amblyopia Treatment Study protocols on patients in this age range, we have found no indication that the response to patching treatment is related to age. Therefore, it is highly unlikely that a delay in initiating treatment of weeks or even months could be harmful.

This study is addressing issues related to the treatment of amblyopia in children 3 to <7 years old with visual acuity 20/40 to 20/400. The study consists of two phases:

1. a Spectacle Phase in which patients are prescribed spectacles and followed until maximal improvement in visual acuity has occurred and
2. a Randomized Trial comparing a group using patching treatment (in addition to spectacle correction) with a control group using spectacle correction only.

The sample size for the primary analysis for the randomized trial has been estimated to be 134 patients. Patients will be enrolled into the Spectacle Phase until the recruitment goal for the Randomized Trial is reached.

ELIGIBILITY:
Inclusion Criteria:

* Age 3 to <7 years
* Able to perform visual acuity using the ATS single-surround HOTV protocol
* Amblyopia associated with strabismus (comitant or incomitant), anisometropia, or both
* Visual acuity in the amblyopic eye 20/40 to 20/400 inclusive
* Visual acuity in the sound eye >20/40
* Inter-eye acuity difference >3 logMAR lines
* Cycloplegic refraction and ocular examination within 2 months prior to enrollment

Exclusion Criteria:

* No amblyopia treatment (other than spectacles) in the past month and no more than one month of amblyopia treatment in the past 6 months
* No current vision therapy or orthoptics
* No ocular cause for reduced visual acuity
* No myopia more than a spherical equivalent of -6.00 D
* No prior intraocular or refractive surgery
* No known skin reactions to patch or bandage adhesives

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 268
Dates: Start 2004-02; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
maximal improvement in visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: David K. Wallace, M.D., Study Chair — Duke University Eye Center; Susan A. Cotter, O.D., Study Chair — Southern California College of Optometry at Marshall B. Ketchum University
Locations (2):
- United States (2):
  - Southern California College of Optometry, Fullerton, California
  - Duke University Eye Center, Durham, North Carolina

REFERENCES:
- [Result] Cotter SA; Pediatric Eye Disease Investigator Group; Edwards AR, Wallace DK, Beck RW, Arnold RW, Astle WF, Barnhardt CN, Birch EE, Donahue SP, Everett DF, Felius J, Holmes JM, Kraker RT, Melia M, Repka MX, Sala NA, Silbert DI, Weise KK. Treatment of anisometropic amblyopia in children with refractive correction. Ophthalmology. 2006 Jun;113(6):895-903. doi: 10.1016/j.ophtha.2006.01.068. PMID 16751032
- [Result] Wallace DK; Pediatric Eye Disease Investigator Group; Edwards AR, Cotter SA, Beck RW, Arnold RW, Astle WF, Barnhardt CN, Birch EE, Donahue SP, Everett DF, Felius J, Holmes JM, Kraker RT, Melia M, Repka MX, Sala NA, Silbert DI, Weise KK. A randomized trial to evaluate 2 hours of daily patching for strabismic and anisometropic amblyopia in children. Ophthalmology. 2006 Jun;113(6):904-12. doi: 10.1016/j.ophtha.2006.01.069. PMID 16751033
- [Derived] Wallace DK, Lazar EL, Melia M, Birch EE, Holmes JM, Hopkins KB, Kraker RT, Kulp MT, Pang Y, Repka MX, Tamkins SM, Weise KK; Pediatric Eye Disease Investigator Group. Stereoacuity in children with anisometropic amblyopia. J AAPOS. 2011 Oct;15(5):455-61. doi: 10.1016/j.jaapos.2011.06.007. PMID 22108357
- [Derived] Repka M, Simons K, Kraker R; Pediatric Eye Disease Investigator Group. Laterality of amblyopia. Am J Ophthalmol. 2010 Aug;150(2):270-4. doi: 10.1016/j.ajo.2010.01.040. Epub 2010 May 8. PMID 20451898
- See also: Pediatric Eye Disease Investigator Group — http://pedig.net